CLINICAL TRIAL: NCT02215304
Title: A Randomized, Double-blind, Placebo-controlled Intervention Study to Assess the Safety and Tolerance Effect of Three Probiotic Strains in Infants
Brief Title: Safety and Tolerance Study of Three Probiotic Strains in Infants
Acronym: PROBINFANT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ProbiSearch SL (Industry)
Collaborators: Lallemand Health Solutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: LALLEM-001
Record Dates: First submitted 2014-08-11; First posted 2014-08-13 (Estimated); Last update posted 2016-12-14 (Estimated); Status verified 2016-12

CONDITIONS: Body Weight; Body Height; Head Circumference
Keywords: Dietary supplementation; Probiotics; Safety/Efficiency; Healthy infants
MeSH Terms: conditions — Body Weight

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Bifidobacterium longum R0033 (Active Comparator): Bifidobacterium longum ssp infantis R0033, 3*10E9 colony forming units (CFU) in 1 sachet per day to be diluted in 10 mL water by mouth for eight weeks
  Interventions: Dietary Supplement: Bifidobacterium longum ssp infantis R0033
- Lactobacillus helveticus R0052 (Active Comparator): Lactobacillus helveticus R0052, 3*10E9 colony forming units (CFU) in 1 sachet per day to be diluted in 10 mL water by mouth for eight weeks
  Interventions: Dietary Supplement: Lactobacillus helveticus R0052
- Bifidobacterium bifidum R0071 (Active Comparator): Bifidobacterium bifidum R0071, 3*10E9 colony forming units (CFU) in 1 sachet per day to be diluted in 10 mL water by mouth for eight weeks
  Interventions: Dietary Supplement: Bifidobacterium bifidum R0071
- Placebo (Placebo Comparator): potato starch 1 sachet per day to be diluted in 10 mL water by mouth for eight weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Bifidobacterium longum ssp infantis R0033 — 12 weeks intervention study: A run-in period of two weeks, 8 weeks of intervention (from weeks 2 to 10) and two weeks after intervention finishing time.
  During the 8 weeks of intervention participants will intake one daily dose of the product which contains 3*10E9 colony forming units (CFU)
  Arms: Bifidobacterium longum R0033
Dietary Supplement: Lactobacillus helveticus R0052 — 12 weeks intervention study: A run-in period of two weeks, 8 weeks of intervention (from weeks 2 to 10) and two weeks after intervention finishing time.
  During the 8 weeks of intervention participants will intake one daily dose of the product which contains 3*10E9 colony forming units (CFU)
  Arms: Lactobacillus helveticus R0052
Dietary Supplement: Bifidobacterium bifidum R0071 — 12 weeks intervention study: A run-in period of two weeks, 8 weeks of intervention (from weeks 2 to 10) and two weeks after intervention finishing time.
  During the 8 weeks of intervention participants will intake one daily dose of the product which contains 3*10E9 colony forming units (CFU)
  Arms: Bifidobacterium bifidum R0071
Dietary Supplement: Placebo — 12 weeks intervention study: A run-in period of two weeks, 8 weeks of intervention (from weeks 2 to 10) and two weeks after intervention finishing time.
  During the 8 weeks of intervention participants will intake one daily dose of the product which contains 3*10E9 colony forming units (CFU)
  Arms: Placebo

SUMMARY:
Study to evaluate the safety and tolerance of three probiotic bacteria intake by healthy infants. Participants are divided at random and unknown to the researchers, in four groups, three of which receive one of three probiotic bacteria while the fourth group receives placebo product.

DETAILED DESCRIPTION:
Subjects' parents or legal tutors will be contacted for voluntary participation and a written informed consent will be obtained.

The study visits will take place either in the hospital or primary health center.

During Visit 1, inclusion in- and exclusion criteria will be checked and information on demographic profile, subject characteristics, feeding option, relevant medical history, medication and nutritional supplements will be recorded. Weight and length and head circumference measurements of the infant will be made. The researcher will explain to the parents that during the first 2 weeks of participation in the study the infant must not intake any probiotic supplements (run-in ). Parents will be instructed to collect and send and/or store fecal and urine samples before starting the study. In addition they will be instructed to collect and send and/or store fecal and urine samples after the initial run-in period (2 weeks), after the product intake period (8 weeks) and after the final wash out period (2 weeks).

During Visit 2, subjects will be randomly allocated to receive either one of the test products or the placebo. Body weight and length will be measure. The researcher will review with the parents the study diary in detail, how to record data on gastrointestinal tolerance, stool frequency and stool characteristics, respiratory symptoms, diagnosed infections, sleeping and crying habits, changes in sleeping pattern, fever episodes, unscheduled visits resulting from suspected infection or a health problem and antibiotic prescription. The researcher will explain the procedure of administering the study product to the infant and anticipated phone calls. The parents will be instructed to start intake of the product as soon as possible after the collection of fecal and urine samples.

During product intake period (8 weeks) subject's parents will be called weekly by someone from the Study Team (Phone call 1, 2, 3, 4, 5, 6, 7). During the phone call relevant data related to possible Adverse Events (AEs) or Serious Adverse Events (SAEs) will be collected. Parents will be asked about infant's well-being (fever episodes, rashes, diarrhea, visits to the doctor, antibiotic prescription, etc.). Issues regarding diary completion, if any, will be discussed. During the Phone call 7 parents will be instructed to collect and send and/or store fecal and urine samples in one of the days prior to the third visit.

At the third visit (Visit 3, 8 weeks after product intake period), body weight and length will be measured and relevant data will be collected with respect to health and well-being aspect of the infant and AE or SAE (fever episodes, rashes, diarrhea, visits to the doctor, antibiotic prescription, etc.). Completed diaries and fecal and urine samples will be collected. Parents will be explained that for the last 2 weeks of participation in the study their infants could not intake any probiotic supplement (final wash out period). Parents will be instructed to collect and send and/or store fecal and urine samples in one of the days prior to the next visit (Visit 4).

During visit 4, after the final wash out period, body weight and length will be measured and relevant data will be collected with respect to health and well-being aspect of the infant and AEs or SAEs (fever episodes, rashes, diarrhea, visits to the doctor, antibiotic prescription, etc.). Completed diaries and samples will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Healthy term infants between 3-12 months old
* Written informed consent from at least one parent or the legal tutor.

Exclusion Criteria:

* Short bowel syndrome or any GI surgery.
* Impaired intestinal epithelial barrier (e.g. diarrheal illness, intestinal inflammation).
* Metabolic disorders (diabetes, lactose intolerance).
* Immunodeficiency.
* Heart failure and cardiac medical history (e.g. artificial heart valve, medical history of infectious endocarditis, cardiac malformation, rheumatic fever).
* Surgery within one month prior to inclusion (Visit 1/ week 0).
* Antibiotic prescription 1 week before inclusion (Visit 1/ week 0) and during run-in period (Visit 2/ week 2).
* Investigator's uncertainty about the willingness or ability of the infant's parents to comply with the protocol requirements.
* Participation in any other clinical trial within two weeks prior to entry into the study.

Ages: 3 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 221 (Actual)
Dates: Start 2014-06; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Safety and tolerance will be evaluated according to infant growth (weight, height and head circumference) | 12 weeks
  growth will be evaluated considering weight, height and head circumference, at four different time points during study: 1st measure will be at screening visit (visit 1/week 0), 2nd measure will be after the run-in period and before starting intervention (visit 2/ week 2), 3rd measure will be after the eight weeks of intervention (visit 3/ week 10) and the 4th measure will be two weeks later (visit 4/week 12).
Adverse Event and/or Serious Adverse Event | 10 weeks
  Adverse Event and/or Serious Adverse Event will be recorded daily by parents and notified to investigator within 24hrs., in particular gastro-intestinal symptoms, fever and rashes.
Fecal characteristics | 10 weeks
  Fecal characteristics (stool frequency, stool consistency, stool amount and stool color) will be recorded daily by parents according to the "Amsterdam scale" and notified weekly to investigators.
Use of medication | 12 weeks
  Medication used (antibiotics, etc) will be recorded daily by parents and notified weekly to investigators.

SECONDARY OUTCOMES:
Urine concentration of D-lactic acid. | 12 weeks
  D-lactic acid will be measured in urine samples at 4 different time points (weeks 0, 2, 10 and 12).
Changes in sleep and crying patterns | 10 weeks
  Changes in sleep and crying patterns will be recorded daily by parents and notified weekly to investigators.
Immune compounds in fecal samples | 8 weeks
  Immunoglobulins (Ig) A, G1, G2, G3, G4 and M, cytokines, chemokines and growth factors such as interleukins (IL) 1β, 2, 4, 5, 6, 7, 8, 10, 12, 13, and 17, interferon-γ (INF-γ), tumor necrosis factor-α (TNF-α), growth related oncogene-α (GRO-α), macrophages chemoattractant protein-1 (MCP-1), macrophages inflammatory protein-1β (MIP-1β), granulocyte-colony stimulating factor (G-CSF), granulocyte-macrophages colony stimulating factor (GM-CSF) and Calprotectin concentrations will be measured at two time points, before and after the study probiotic intake (weeks 0 and 10).
Composition of fecal microbiota | 8 weeks
  Composition of fecal microbiota will be assessed at two different time points, before and after the intervention period

CONTACTS AND LOCATIONS:
Overall Officials: Felix Omeñaca, MD, PhD, Principal Investigator — Hospital Universitario La Paz
Locations (1):
- Hospital Universitario La Paz, Madrid, Madrid, Spain